CLINICAL TRIAL: NCT03059199
Title: HAT TRICK: Examining the Feasibility of a Gender Sensitive Intervention Focused on Physical Activity, Healthy Eating and Connectedness in Male Hockey Fans
Brief Title: HAT TRICK: An Innovative Health Promotion Program for Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Cristina Caperchione, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H1600736
Record Dates: First submitted 2016-11-18; First posted 2017-02-23 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Cancer Prevention
Keywords: Prospective/Retrospective

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-Arm Feasibility Study (Experimental): 12-week, 1x/week, 90-minute face-to-face sessions.
  Interventions: Behavioral: Single-Arm Feasibility Study

INTERVENTIONS:
Behavioral: Single-Arm Feasibility Study — Participants are provided with the HAT TRICK Playbook, a resource manual including weekly healthy eating and physical activity challenges and tracking logs. Each face-to-face session is facilitated by trained research staff, community partners, and health care professionals. Weekly sessions include information on physical activity, healthy eating, and behaviour change techniques (e.g., social support, goal setting, self-monitoring) and include an opportunity to be active/exercise.

SUMMARY:
The purpose of this research is to implement and evaluate the feasibility of the HAT- TRICK Program, a gender- sensitive intervention program targeting physical activity, healthy eating and connectedness in men living in the Okanagan Region, BC.

DETAILED DESCRIPTION:
Despite the benefits associated with lifestyle changes, men are less likely than women to engage in healthy lifestyle behaviours. Many men are reluctant and/or 'hard-to-reach', making it difficult to implement chronic illness prevention initiatives. Traditionally, a central challenge associated with engaging men in their health were perceptions that attention to one's health ran counter to masculine ideals of strength, self-reliance and independence. Thus, many men refrain from engaging in health promotion behaviors, such as PA and healthy eating. Research has highlighted the potential for professional sports teams/clubs to attract and engage men in healthy lifestyle behaviours. Such a strategy has been recognised as very powerful due to the traditional male environment within these clubs and the social-cultural connections the men often make with particular teams in terms of loyalty, identity and belonging. Thus, the purpose of this research is to develop and evaluate the feasibility of the HAT-TRICK Program, a gender-sensitive intervention program targeting PA, healthy eating and connectedness in men living in Kelowna, BC. This program will be delivered as a collaborative effort between the research team and the Kelowna Rockets, a major junior ice hockey team in Kelowna, BC. The Kelowna Rockets play in a centre with a capacity of over 6,000 and have one of the most loyal season ticket holders base in the Western Hockey League, with 4,500; the majority being men and between the ages of 40-70 years old. With assistance from the Rockets, participants (N=30) will be recruited via season ticket holders, at hockey games, though the Rockets webpage and local print and electronic media. Participants meeting all eligibility criteria will be invited to participate in the 12 week HAT-TRICK Program which will consist of a once a week, 90 minute combined physical activity (e.g., resistance training, "boot-camp" training, floor hockey, stair climbing) and health education session (e.g., goal setting, self-monitoring, barriers and benefits to PA, dealing with set-backs, healthy eating, alcohol consumption, etc.) to be held at the Kelowna Rockets game and training facility. Kelowna Rockets personnel (e.g., athletic therapist, nutritionist) and community experts (e.g., chef, fitness trainer) will be invited to lead some of the PA and nutrition sessions. Kelowna Rockets players will also visit the group during selected sessions to engage in the PA training with the men, further encouraging social support, connectedness and camaraderie. Primary (feasibility and acceptability) and secondary (PA, nutrition, quality of life, connectedness, anthropometrics) outcome measures will be evaluated using a mix-methods approach including; focus groups, self-reported questionnaires and objective physical activity and anthropometric methods. All measures will be collected at baseline, post-intervention (12 weeks) and at 9-month follow-up. Findings from the primary and secondary outcome measures will be used to refine the HAT-TRICK program in preparation for a full-scale evaluation (RCT). Innovative prevention and health promoting approaches are needed to better serve this 'hard to reach' population. This innovative program utilizes a gender sensitive approach to attract and engage men, providing them with a program that recognises their masculine values and interests. Furthermore, the collaborative (i.e., Kelowna Rockets) nature of this program is poised to reach a large proportion of men in the Okanagan by capitalizing on the social-cultural connections men often make with sports teams and using this as the lynchpin to engaging men in health behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 35 years
* Residing in the Okanagan Region of British Columbia Canada
* Accumulate <150mins of moderate to vigorous physical activity a week
* Have a BMI >25kg/m2
* Pant size of >38"

Exclusion Criteria:

* No specific exclusion criteria

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Program Feasibility | Post-Intervention (12-weeks)
  Program feasibility will be evaluated using mixed-methods to explore program delivery, recruitment, participant and facilitator satisfaction, challenges and issues faced during the program, and recommended changes to the program. Methods for collecting feasibility data will include: 1) program satisfaction/acceptability questionnaire for all participants; 2) semi-structured telephone interviews with a sub-sample of the HAT TRICK participant (telephone interviews provide rich qualitative data and are time & resource efficient; 3) semi-structured interviews with guest presenters and club 'insiders'.

SECONDARY OUTCOMES:
Dietary Behaviour | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measured by the Dietary Instrument for Nutrition Education (DINE) questionnaire.
Physical Activity Behaviour | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measured using the Actigraph GT3X+© accelerometer and Godin's Leisure Time Exercise Questionnaire (GLTEQ). The Actigraph GT3X+©, which is the 'gold standard' measure of physical activity in adults, will be worn by all participants during all waking hours over 7 consecutive days.
Anthropometrics | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measures of height, weight, waist circumference, and blood pressure
Health-Related Quality of Life | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Health-related quality of life will be assessed using the validated SF-12V2 Health Survey.
Social Connectedness | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measured using the Abbreviated Duke Social Support Scale.
Alcohol Consumption | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measured using a 7-day alcohol recall.
Sedentary Behaviour | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measured using the Marshall Sitting Questionnaire.
Risk of Depression | Baseline, Post-Intervention (12-weeks), and 9-month follow-up
  Measured using the Male Depression Risk Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Caperchione, PhD, Principal Investigator — UBCO Health and Exercise Sciences
Locations (1):
- Prospera Place, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Only the principal investigators and UBC research team members will have access to the raw data. CO-I's external to UBC will not require access to raw participant data. Any data that are shared will be aggregate data and have all identifiers removed. All of these individuals have training in issues concerning privacy, confidentiality, and are aware of their responsibilities to maintain these.

REFERENCES:
- [Background] Caperchione CM, Bottorff JL, Oliffe JL, Johnson ST, Hunt K, Sharp P, Fitzpatrick KM, Price R, Goldenberg SL. The HAT TRICK programme for improving physical activity, healthy eating and connectedness among overweight, inactive men: study protocol of a pragmatic feasibility trial. BMJ Open. 2017 Sep 6;7(9):e016940. doi: 10.1136/bmjopen-2017-016940. PMID 28882920
- [Result] Sharp P, Bottorff JL, Hunt K, Oliffe JL, Johnson ST, Dudley L, Caperchione CM. Men's Perspectives of a Gender-Sensitized Health Promotion Program Targeting Healthy Eating, Active Living, and Social Connectedness. Am J Mens Health. 2018 Nov;12(6):2157-2166. doi: 10.1177/1557988318799159. Epub 2018 Sep 20. PMID 30234419
- [Derived] Sharp P, Bottorff JL, Oliffe JL, Hunt K, Caperchione CM. Process evaluation of HAT TRICK: feasibility, acceptability and opportunities for programme refinement. Health Educ Res. 2020 Dec 23;35(6):605-617. doi: 10.1093/her/cyaa029. PMID 33099636
- See also: HAT TRICK program information and participant recruitment webpage — http://www.hattrick.ok.ubc.ca